CLINICAL TRIAL: NCT06605846
Title: Otago Exercises on the Risk of Falling in Prostatic Cancer Patients Receiving Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, lectrurer of physical therapy for general surgery, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005337
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Prostate
Keywords: Androgen deprivation therapy; otago excercises; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercise training (Experimental): This group included 52 patients receive Otago exercise training for 45 minutes after each session with routine medical care for prostatic cancer patients
  Interventions: Other: otago excercises
- control (Sham Comparator): This group included 52 patients receive routine medical care for prostatic cancer patients.
  Interventions: Other: Medical ADT treatment

INTERVENTIONS:
Other: otago excercises — Otago training is helpful, and one of the most powerful interventions where the original randomized controlled trials reported improvements in functional outcomes and a 35% reduction in falls for frail, high-risk older adults (Shubert et al., 2018). In Egypt, there are little researches about Otago Exercise Program.
  Exercise is well-known as an economic and key adjuvant treatment in clinical oncology that improves QOL of cancer survivors. Many studies focused on investigating the benefits of exercise interventions on preventing falls and improving physical performance of older adults. Combination of strength and functional balance exercise has been demonstrated as an effective method to improve balance performance, rather than strength training alone
  Arms: Otago exercise training
Other: Medical ADT treatment — Medical ADT treatment according to patient age, prostatic cancer stage
  Other Names: control
  Arms: control

SUMMARY:
Androgen deprivation therapy (ADT) is a common treatment for older men with advanced prostate cancer (PCa) but is associated with numerous deleterious health effects that may accentuate age associated physiological declines.

Decreased lower body muscle mass and strength, cognitive decline, worsen fatigue and progressive loss of BMD following initiating ADT could put prostate cancer survivors at higher risk of impaired physical functioning performance and subsequently developing falls. Otago training is helpful, and one of the most powerful interventions where the original randomized controlled trials reported improvements in functional outcomes and a 35% reduction in falls for frail, high-risk older adults (Shubert et al., 2018). In Egypt, there are little researches about Otago Exercise Program.

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) is a common treatment for older men with advanced prostate cancer (PCa) but is associated with numerous deleterious health effects that may accentuate age associated physiological declines.

Decreased lower body muscle mass and strength, cognitive decline, worsen fatigue and progressive loss of BMD following initiating ADT could put prostate cancer survivors at higher risk of impaired physical functioning performance and subsequently developing falls.

Otago training is helpful, and one of the most powerful interventions where the original randomized controlled trials reported improvements in functional outcomes and a 35% reduction in falls for frail, high-risk older adults (Shubert et al., 2018). In Egypt, there are little researches about Otago Exercise Program.

Exercise is well-known as an economic and key adjuvant treatment in clinical oncology that improves QOL of cancer survivors. Many studies focused on investigating the benefits of exercise interventions on preventing falls and improving physical performance of older adults. Combination of strength and functional balance exercise has been demonstrated as an effective method to improve balance performance, rather than strength training alone

ELIGIBILITY:
Inclusion Criteria:

* Men aged 50 years or older diagnosed with adenocarcinoma prostate cancer.

  * Will initiate and receive continuous ADT (luteinizing hormone releasing hormone agonist (LHRH) or combination of LHRH and anti-androgen) for at least 6 months after recruitment.
  * Report > 1 fall in the past year OR have a score on one of two physical performance tests that is associated with increased fall risk (i.e., ≥ 12.0 s to complete the 3 m timed up and go (TUG)
  * Willing to attend >75% of intervention Otago exercises

Exclusion Criteria:

* severe cardiac disease (New York Heart Association class III or greater), angina,
* uncontrolled hypertension (blood pressure > 160/95 mmHg), moderate to severe aortic stenosis, acute illness or fever, uncontrolled atrial or ventricular dysrhythmias, uncontrolled sinus tachycardia (> 120 beats per minute), third-degree atrioventricular heart block
* lower limb fracture within last 3 months , lower limb amputation

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Isometric knee muscle strength | base line and 24 weeks
  will be used to evaluate knee extension and flexion isometric strength.
Bone mineral density (BMD | base line and 24 weeks
  will be used to evaluate Bone mineral density of the lumbar spine (LS) and femoral neck (FN)

SECONDARY OUTCOMES:
Timed up and go (TUG) test | base line and 24weeks
  will be used to measure basic mobility skills. The measurement outcome for TUG is the time it takes to rise up out of a chair, walk 3 m away from the chair, walk 3 m back to the chair, and return to the seated position
Berg Balance Scale (BBS) | base line and 24weeks
  Used to assess the patient ability to balance his /her body during activities and risk of fall

CONTACTS AND LOCATIONS:
Locations (1):
- MTI university, Multiple Locations, Egypt

IPD SHARING:
Plan to Share IPD: No